CLINICAL TRIAL: NCT07250087
Title: Phase 1 Study of Asciminib Maintenance Therapy Following Allogeneic Stem Cell Transplant or Chimeric Antigen Receptor T Cell Therapy (CAR T) to Prevent Relapse in Adults With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Brief Title: Asciminib Maintenance Therapy Following alloHCT or CAR T to Prevent Relapse in Adults With Ph+ALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23477
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
MeSH Terms: interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients post-alloHCT (Experimental): Individuals who have previously undergone an allogeneic stem cell transplant (alloHCT).
  Interventions: Drug: Asciminib
- Patients post-CAR T cell therapy (Experimental): Individuals who have received chimeric antigen receptor T cell therapy (CAR T).
  Interventions: Drug: Asciminib

INTERVENTIONS:
Drug: Asciminib — Treatment will be administered on an outpatient basis.

SUMMARY:
The purpose of the study is to see if a study drug called asciminib is safe and okay for people to take after they've had treatment for a type of blood cancer called Philadelphia Chromosome

Positive Acute Lymphoblastic Leukemia (Ph+ B-ALL). We're looking at two groups of adults:

one group had an Allogeneic Stem Cell Transplant (alloHCT) cohort A, and the other group had chimeric antigen receptor T cell (CAR T) therapy, cohort B. We also want to figure out what the best dose of asciminib is to use moving forward in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of Ph+ B-ALL with detectable Philadelphia chromosome abnormalities
* Morphologic remission (<5% marrow blasts)
* ECOG performance status 0-2
* Adequate organ function

Exclusion Criteria:

* Active relapsed disease (>5% blasts)
* Grade II-IV acute GVHD requiring systemic steroids
* Significant organ dysfunction or uncontrolled infection
* Pregnancy or breastfeeding
* Prior investigational CAR T product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose | Up to 24 months
  The MTD is defined as the highest dose level at which one or none of six patients experience a DLT.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | Up to 24 Months
  Relapse-free survival (RFS) is defined as the time from starting asciminib to the date of relapse or death, whichever comes first.
Overall survival (OS) | Up to 24 Months
  Overall survival (OS) is defined as the time from starting asciminib to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Rawan Faramand, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States